CLINICAL TRIAL: NCT01630564
Title: Phase I Study of Ex Vivo Expanded Donor Cord Blood T-Lymphocyte Infusion in Post-Transplant Relapsed Patients
Brief Title: Donor Cord Blood T-Cell Infusion After Stem Cell Transplant in Treating Patients With Relapsed Hematological Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1178; NCI-2013-00385 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-1178 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (T-cell infusion) (Experimental): Patients undergo ex vivo-expanded umbilical cord blood progenitor cell donor T cell infusion with aldesleukin 11-14 days after T-cell co-stimulation begins.
  Interventions: Biological: Aldesleukin; Procedure: Ex Vivo-Expanded Cord Blood Progenitor Cell Infusion; Biological: Umbilical Cord Blood-Derived Lymphocyte Therapy

INTERVENTIONS:
Biological: Aldesleukin — Undergo ex-vivo-expanded umbilical cord blood progenitor cell donor T-cell infusion with aldesleukin
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Procedure: Ex Vivo-Expanded Cord Blood Progenitor Cell Infusion — Undergo ex-vivo-expanded umbilical cord blood progenitor cell donor T-cell infusion with aldesleukin
Biological: Umbilical Cord Blood-Derived Lymphocyte Therapy — Undergo ex-vivo-expanded umbilical cord blood progenitor cell donor T-cell infusion with aldesleukin

SUMMARY:
This phase I trial studies the side effects and best dose of donor cord blood T-cells after stem cell transplant in treating patients with relapsed hematological malignancies. After umbilical cord blood transplant, stem cells are collected from the donor's cord blood and stored. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by treatment. Removing the T cells and treating them in the laboratory before infusing them in the patient may also help boost the patient's immune system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and maximum tolerated dose (MTD) of infusion of ex vivo expanded cord blood T cells (CLI), in cord blood (CB) transplant recipients with relapsed hematological malignancies.

SECONDARY OBJECTIVES:

I. To determine the complete remission rate and overall response as a result of CLI infusion.

II. To determine the effect of CLI infusion on the chimerism. III. To evaluate the incidence rate and grade of acute graft-versus-host disease (GvHD) after CLI infusion.

IV. To determine the disease-free survival, cytopenia rate, relapse incidence after CLI infusion.

OUTLINE: This is a dose-escalation study of ex vivo-expanded T-cells.

Patients undergo ex vivo-expanded umbilical cord blood progenitor cell donor T cell infusion with aldesleukin 11-14 days after T-cell co-stimulation begins.

After completion of study treatment, patients are followed up for 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Umbilical cord blood (UCB) recipients with underlying hematological malignancies presenting with post-transplant relapse and have available approximately 400 microliter to 1 ml aliquots or CB wash from previous transplant
* UCB recipients with T-cell and/or overall chimerism value of less than 80%, in absence of relapse and have available approximately 400 microliter to 1 ml aliquots or CB wash from previous transplant
* Performance score of at least 80% by Karnofsky or performance status (PS) < 3 (Eastern Cooperative Oncology Group [ECOG]) (age >= 12 years), or Lansky Play-performance scale of at least 60% or greater (age < 12 years)
* Negative beta human chorionic gonadotropin (HCG) or urine test in females of childbearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization and willing to use an effective contraceptive measure while on the study
* Patient or patient's legal representative, parent(s) or guardian able to sign informed consent

Exclusion Criteria:

* Human immunodeficiency virus (HIV) positive (due to the extreme immunosuppressive nature of allogeneic stem cell transplant)
* Patients with active (untreated) central nervous system (CNS) disease
* Any active GVHD
* Active invasive infections
* Pregnant or breast-feeding

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-03-11 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ex vivo expanded T-cells defined as the highest dose for which the probability of toxicity is closest to 30% without exceeding 30% | Up to day 45
  Dose limiting toxicity is defined as grade IV graft-versus-host disease (GVHD), grades 3-4 acute GVHD occurring within 45 days of the study T cell infusion, grade 3-5 organ toxicity (cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic), grade 4 cytopenia, or any grade 4 or 5 organ based (non-hematologic) toxicity.

SECONDARY OUTCOMES:
Incidence of adverse events by grade by ex vivo expanded cord blood T cells dose and overall | Up to day 100
Numbers of patients treated at the MTD with grade 2-4 GVHD | Up to day 100
  Estimated with an exact 95% binomial confidence interval.
Proportion of patients with remission post-infusion | Up to day 100
  Estimated with an exact 95% binomial confidence interval.
Proportion of patients achieving chimerism post-infusion | Up to day 100
  Estimated with an exact 95% binomial confidence interval.
Proportion of patients with cytopenia post-infusion | Up to day 100
  Estimated with an exact 95% binomial confidence interval.
Proportion of patients that relapse after infusion | Up to day 100
  Estimated with an exact 95% binomial confidence interval.
Disease-free survival | Up to day 100
  Estimated with the Kaplan-Meier product limit estimator.

CONTACTS AND LOCATIONS:
Overall Officials: Sairah Ahmed, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org